CLINICAL TRIAL: NCT06930430
Title: Gingival Crevicular Fluid Sphingosine-1-phosphate and Interleukin-1 Beta Levels After Non-surgical Periodontal Therapy: a Split-mouth Randomized Trial
Brief Title: IL-1β and S1P Levels After Periodontal Therapy: A Split-Mouth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Atanur Sarioglu, Research assistant, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMU KAEK protokol no: 2023/96
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sphingosine 1-phosphate; Interleukin 1-beta; Gingival Crevicular Fluid; Non-surgical Periodontal Therapy; Split-mouth Design
Keywords: gingival crevicular fluid; sphingosine-1-phosphate; interleukin-1 beta; non-surgical periodontal therapy

STUDY DESIGN:
Intervention Model Description: This study followed a single group, split-mouth design. Seventeen systemically healthy, non-smoking patients with stage III periodontitis were included. For each participant, three periodontally diseased sites (with PD ≥ 6 mm and CAL ≥ 5 mm) and three periodontally healthy control sites (with PD ≤ 3 mm and no CAL) were selected. This resulted in a total of 51 diseased and 51 healthy sites for comparative evaluation. All patients received full-mouth non-surgical periodontal therapy. Biochemical and clinical outcomes were assessed longitudinally at baseline, 1 month, and 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stage III Periodontitis Patients (Other): This arm included 17 systemically healthy, non-smoking patients diagnosed with stage III periodontitis. Each participant contributed three periodontally diseased sites and three periodontally healthy sites, resulting in a total of 51 diseased and 51 healthy sites for evaluation. All patients received full-mouth non-surgical periodontal therapy. Clinical and biochemical parameters were assessed at baseline, 1 month, and 3 months.
  Interventions: Procedure: Non-Surgical Periodontal Therapy (NSPT)

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Therapy (NSPT) — Scaling and root planing was performed using hand instruments under local anesthesia, if necessary. Oral hygiene instructions were provided using the modified Bass technique. GCF samples were collected from the same sites at baseline, 1 month, and 3 months to measure levels of IL-1β and S1P using ELISA.

SUMMARY:
This randomized split-mouth clinical trial aimed to evaluate the changes in interleukin-1 beta (IL-1β) and sphingosine-1-phosphate (S1P) levels in gingival crevicular fluid (GCF) following non-surgical periodontal therapy (NSPT) in patients with stage III periodontitis. A total of 17 systemically healthy, non-smoking individuals were included. For each patient, three diseased and three healthy periodontal sites were selected, totaling 51 diseased and 51 healthy sites for biochemical and clinical evaluation.

GCF samples and clinical periodontal parameters were collected at baseline, one month, and three months after NSPT. The levels of IL-1β and S1P were quantified using enzyme-linked immunosorbent assay (ELISA). The study also investigated the correlation between biomarker levels and clinical indicators of periodontal disease severity, such as probing depth and clinical attachment level.

DETAILED DESCRIPTION:
Diseased sites were selected based on the most severe clinical findings, including probing depth (PD) of ≥6 mm, clinical attachment level (CAL) of ≥5 mm, and the presence of bleeding on probing (BOP). Healthy sites were defined by PD ≤3 mm, no clinical attachment loss, absence of radiographic bone loss, and BOP negativity. All selected sites were non-adjacent and distributed throughout the oral cavity to reduce regional bias.

This study also aimed to explore site-specific changes in biomarker expression over time and assess the correlation between GCF IL-1β/S1P levels and clinical indicators of periodontal disease severity and healing response. All GCF sampling was repeated from the same sites at each time point. Control (healthy) site sampling was done at baseline and 3 months, while diseased site sampling was conducted at baseline, 1 month, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45 and 60 years
* Systemically healthy individuals with no known systemic conditions
* Non-smokers or former smokers who had quit at least two years prior
* Diagnosed with Stage III periodontitis according to the 2017 World Workshop Classification
* Presence of at least three diseased sites with probing depth (PD) ≥ 6 mm, clinical attachment level (CAL) ≥ 5 mm, and bleeding on probing (BOP [+])
* Presence of at least three periodontally healthy sites with PD ≤ 3 mm, no CAL, and no BOP
* No periodontal treatment within the last 6 months
* Provided written informed consent

Exclusion Criteria:

* Presence of systemic diseases known to affect periodontal status (e.g., diabetes mellitus, cardiovascular disease, autoimmune disorders)
* Use of antibiotics or anti-inflammatory medications within the last 6 months
* History of periodontal surgery within the past 12 months
* Pregnant or lactating women
* Current smokers or individuals who quit less than two years ago
* Sites with endodontic lesions, caries extending to the cervical area, trauma-related gingival recession, or bone loss due to non-periodontal causes
* Undergoing orthodontic treatment during the study period

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in gingival crevicular fluid (GCF) sphingosine-1-phosphate (S1P) levels | Baseline, 1 month, and 3 months
  S1P levels in gingival crevicular fluid (GCF) were measured using ELISA at diseased and periodontally healthy sites. Changes were evaluated at baseline, 1 month, and 3 months following non-surgical periodontal therapy (NSPT).
Change in gingival crevicular fluid (GCF) interleukin-1 beta (IL-1β) levels | Baseline, 1 month, and 3 months
  IL-1β levels in gingival crevicular fluid (GCF) were quantified via ELISA at both diseased and periodontally healthy sites. Changes were evaluated at baseline, 1 month, and 3 months following non-surgical periodontal therapy (NSPT).

SECONDARY OUTCOMES:
Correlation between IL-1β and S1P levels in gingival crevicular fluid (GCF) | Baseline, and 3 months
  The study evaluated the statistical correlation between IL-1β and S1P concentrations in gingival crevicular fluid (GCF) samples collected from diseased and periodontally healthy sites at baseline and 3 months after non-surgical periodontal therapy (NSPT).
Correlation of S1P and IL-1β levels with clinical periodontal parameters | Baseline, and 3 months
  The levels of S1P and IL-1β in gingival crevicular fluid (GCF) were analyzed for correlation with clinical periodontal indices, including plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL), and GCF volume. Correlations were evaluated at baseline and 3 months following non-surgical periodontal therapy (NSPT) to assess the association between inflammatory biomarkers and clinical disease activity.
Change in clinical periodontal parameters following non-surgical periodontal therapy (NSPT) | Baseline, 1 month, and 3 months
  Plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL), and GCF volume were recorded at diseased and healthy sites to assess periodontal status. These parameters were evaluated at baseline, 1 month, and 3 months after treatment to monitor clinical response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Atanur Sarioglu, DDS, Principal Investigator — Ondokuz Mayıs University, Department of Periodontology
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No